CLINICAL TRIAL: NCT03801330
Title: Inspiration Point-A Digital Pulmonary Rehabilitation Tool for Use With Self- Management Interventions
Brief Title: Inspiration Point-A Digital Pulmonary Rehabilitation Tool Management Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blue Marble Rehab Inc (Industry)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HL137502
Record Dates: First submitted 2017-08-09; First posted 2019-01-11 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: COPD
Keywords: pulmonary rehabilitation; digital; telehealth; software; electronic health
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Participants in the Usual Care Pulmonary Rehabilitation will receive usual care pulmonary rehab program. Usual care programs typically consist of exercises including upper extremity strengthening, lower extremity strengthening, aerobic exercises such as walking and balance training. Each program is personalized as per the participant's ability. The intervention is usual care exercise and education, which is personalized for each participant. No drugs are being tested in this study.
  Interventions: Other: Usual Care Pulmonary Rehabilitation Program
- Software Tool (Experimental): Participants in the Pulmonary Rehabilitation Software-Based Home Program will use a digital software tool (APP) to obtain the pulmonary rehab home program. Home programs typically consist of exercises including upper extremity strengthening, lower extremity strengthening, aerobic exercises such as walking and balance training. Each program is personalized as per the participant's ability. The intervention is exercise and education, which is personalized for each participant. No drugs are being tested in this study.
  Interventions: Other: Pulmonary Rehabilitation Software-Based Home Program

INTERVENTIONS:
Other: Usual Care Pulmonary Rehabilitation Program — Participants in the Usual Care Pulmonary Rehabilitation Program group will complete an 8 week clinic based Pulmonary Rehabilitation Program (usual care).
  Arms: Usual Care
Other: Pulmonary Rehabilitation Software-Based Home Program — Participants in the Pulmonary Rehabilitation Software-Based Home Program group will complete an 8-week home-based Pulmonary Rehabilitation Program using a software app (software)
  Arms: Software Tool

SUMMARY:
The purpose of this study is to measure the feasibility of use of a digital pulmonary rehabilitation tool compared with standard care home program pulmonary rehabilitation.

DETAILED DESCRIPTION:
The study design is a between subjects (Usual care/App) repeated measures (pre/post) design to compare the feasibility of usual care compared with the digital app, Inspiration Point, used in the home for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have physician permission and diagnosis COPD (FEV1 >30%-80%),
* Gold level A-D, and
* Ability to perform the 6 Minute Walk Test (6MWT).
* This means that participants must meet the standard definition of COPD and have a post-bronchodilator measurement of FEV1/FVC < 0.7.
* All COPD Assessment Test scores will be accepted.
* Patients must have an mMRC score = 1-4.
* Additionally, patients must have taken a Pulmonary Function Test within 1 year or they must retake (for baseline measurement) before participating in the study.
* Patients must not have had a Pulmonary Rehabilitation class within the last 6 months.
* If participants have had a recent cardiac event within 6 months (such as a myocardial infarction or an abnormal cardiac catheterization) they must obtain cardiologist approval before participating in the study.
* In an effort to evaluate feasibility we will request that participants have their own Wi-Fi. Participants may use their own mobile device if they prefer but Blue Marble will have ample supply to provide to participants a device for the purposes of this study.
* Target representativeness for gender, based on COPD demography will be ~50% women, based on recent trends indicating that women have an equal, and perhaps slightly greater risk of COPD compared to men3.
* The Ethnicity/Race target recruitment, consistent with the US and the population at each site.
* Participants must speak, read, and understand English at or above the 6th-grade level (as indicated by having a driver's license or self-report of completion of some high school).

Exclusion Criteria for participants with COPD:

* Pulmonary functional fitness that precludes participation in outpatient/home PR program (i.e. requires in-patient supervision or severity of a co-morbidity that represents a contradiction to exercise in a self-directed program) will be exclusionary.
* A participant who desaturates below SaO2 <88% during the pre-test 6MWT and does not have personal oxygen available will be referred for further evaluation and can be included once they have an O2 titration and supplemental oxygen.
* Other exclusions include if a patient's oxygen use exceeds 4 liters per minute (LPM) or those who score less than 100 meters during the entry 6-minute walk distance.
* Participants with coronary problems will be excluded based on specific morbidity and severity. These coronary exclusions include coronary artery disease with unstable angina.
* Additional exclusions include: any respiratory disorder other than COPD that contraindicates participation in a home-based program.
* The inability to learn how to use Inspiration Point
* An acute neurological or cardiovascular condition such as stroke or acute heart surgery.
* Active cancer with an anticipated survival of less than 6 months or treatment that will preclude them from participating in Pulmonary Rehab.
* A participant with high fall risk as per physician determination.
* The presence of a neurologic disorder that precludes a potential participant from following a typical COPD exercise program or demonstrating hand function sufficient to interface with the tablet.
* This also includes patients with prior or current neurologic event/condition presenting fall risk or requiring assist device for ambulation will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | Change from baseline 6 Minute Walk Test score at 2 months
  Measures distance walked in 6 minutes

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Scale (mMRC) | Change from baseline Modified Medical Research Council Dyspnea Scale (mMRC) score at 2 months
  Single question questionnaire describing shortness of breath. Total Score Range from 0-4, 0 is better.
Medical Outcomes Scale VR-12 | Change from baseline VR-12 score at 2 months
  Survey of health status and quality of life
  From (https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/scoring.html) "Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key given in Table 1. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Table 2 lists the items averaged together to create each scale. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered."
St Georges Respiratory Questionnaire (SGRQ) | Change from baseline St Georges Questionnaire score at 2 months
  A self-administered disease-specific instrument designed to measure the impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. The questionnaire has 50 items Scores range from 0-100, with higher scores indicating more limitations
  https://www.thoracic.org/members/assemblies/assemblies/srn/questionaires/sgrq.php
Lung Information Needs Questionnaire (LINQ) | Change from baseline Lung Information Needs Questionnaire score at 2 months
  The questionnaire used to identify a person with COPD's need for information about their disease. The questionnaire measures the extent to which the patient needs more information, as perceived by the patient and clinician. It is scored to produce an overall score and 6 domain scores (Disease knowledge, medicines, self-management, exercise, diet, smoking).
  The score is the sum of all 6 domains with a range from 0-25. High scores indicate high information needs, a lower score is better.
Software Usability Scale (SUS) | Change from baseline Software Usability Scale (SUS)score at 2 months
  Measures usability and learnability of software tools. Total Score provides percentile score indicating usability/learnability. Range 0-100, Higher (100%) is better.
Timed Up and Go Test (TUG) | Change from baseline TUG score at 2 months
  Measures the time taken to stand up from a chair, walk 10 feet, turn around, and return to sitting.
30 Second Sit to Stand Test (30STST) | Change from baseline 30STST score at 2 months
  Measures the number of times a participant can stand from a seated position in 30 seconds
4 Stage Balance Test (4SBT) | Change in 4STBT score at 2 months
  Measures balance in 4 increasing more challenging positions
COPD Assessment Test (CAT) | Change in CAT score at 2 months
  An 8 item test which measures the effect of COPD on a patient's overall health. The items on this test measure a patient's cough, sputum, breathlessness, chest tightness, confidence, activity, sleep and energy levels
Depression Screen (DS) | Change in DS score at 2 months
  A 2 question survey which can be used to evaluate your risk of depression
Charlson Index (CCI) | Change in CCI score at 2 months
  The Charlson comorbidity index predicts the one-year mortality for a patient who may have a range of comorbid conditions, such as heart disease or cancer (a total of 22 conditions). This index is helpful to ensure the groups are equal for the study comparison and statistics.
Fall Risk Questionnaire (FRQ) | Change in FRQ score at 2 months
  The FRQ is comprised of 13 questions about a person's history of falls and potential fall risk.
Positive Affect and Well-Being Short Form (PROMIS) | Change in PROMIS score at 2 months
  This test is a health-related quality of life questionnaire.
Single Item Literacy Screener (SILS) | Change in SILS score at 2 months
  The SILS is a single item survey which determines literacy and health literacy. It is a direct assessment of a patient's need for assistance in reading health materials.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Flynn, PT PhD, Principal Investigator — Blue Marble Health
Locations (4):
- United States (4):
  - Wake Forest Baptist Health, Charlotte, North Carolina
  - Duke University Healthcare, Durham, North Carolina
  - Cabin Creek Health Systems Inc, Dawes, West Virginia
  - New River Health Association, Scarbro, West Virginia

IPD SHARING:
Plan to Share IPD: No
To be determined